CLINICAL TRIAL: NCT03436602
Title: Multilayer Model for Personalized Risk Stratification of Follicular Lymphoma Patients
Brief Title: Personalized Risk Stratification Model of Follicular Lymphoma Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Oncology Institute of Southern Switzerland (Other)
Collaborators: Azienda Ospedaliero Universitaria Maggiore della Carita (Other); Azienda USL Reggio Emilia - IRCCS (Other Government); Institute of Pathology, Locarno, Ticino, Switzerland (Unknown)
Responsible Party: Sponsor
Other Study IDs: IOSI-EMA-004
Record Dates: First submitted 2018-02-06; First posted 2018-02-19 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Follicular Lymphoma
Keywords: Personalized risk assessment; Risk stratification model
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — FFPE tissue specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training cohort: Cohort of follicular lymphoma patients for the development of the multilayer risk stratification model
- Validation cohort: Cohort of follicular lymphoma patients for the validation of the developed multilayer risk stratification model

SUMMARY:
The study aims at developping and validating an integrated clinico-molecular model for an accurate identification of FL patients who are progression free and progressed, respectively, at 24 months after treatment.

DETAILED DESCRIPTION:
Already existing and coded tumor biological material and health-related personal data will be retrospectively collected. FL diagnosis will be confirmed by central pathology review. Tumor somatic mutations, immunoglobulin gene rearrangement and mutation status will be analyzed by targeted deep next generation sequencing of tumor genomic DNA. Gene expression profiling will be performed by targeted RNA-Seq of biopsy-derived RNA.

An immunohistochemistry panel assessing both tumor phenotype and microenvironment cellular composition will be assessed by Tissue macroarray. FISH will be performed to characterize the most recurrent follicular lymphoma chromosomal translocations.

The adjusted association between exposure variables and progression free survival will be estimated by Cox regression. This approach will provide the covariates independently associated with progression free survival that will be utilized in the development of a hierarchical molecular model to predict progression free survival at 24 months. The hierarchical order of relevance in predicting 24 months progression free survival among covariates will be established by recursive partitioning analysis. Overall, this approach will allow the development of a multilayer dynamic model for anticipating progression within 24 months from treatment.

The model developed in the training set will be tested in the validation sets and the model performance (c-index and net reclassification improvement) in the validation set will be compared with that in the training set. The accuracy of the multilayer model in predicting progression free survival at 24 months will be compared against the FLIPI using c-index and net reclassification improvement.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of FL after January 1st, 2004 (chemoimmunotherapy era)
* Availability of tumor material collected before initiation of medical therapy
* Availability of the baseline and follow-up annotations

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Follicular lymphoma patients
Sampling Method: Probability Sample
Enrollment: 370 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of multilayer personalized stratification model | 24 months after first line treatment
  Assessment of multilayer personalized stratification model accuracy in the identification of patients who are progression free at 24 months after first line therapy plus the proportion of patients correctly identified as progressed within 24 months after first line therapy

SECONDARY OUTCOMES:
Progression free survival | From treatment start to progression / death / last follow-up, up to 13 years of follow-up
  Time elapsed from treatment start to progression (event), death (event) or last follow-up (censoring)
Overall survival | From treatment start to death / last follow-up, up to 13 years of follow-up
  Time elapsed from treatment start to death (event) or last follow-up (censoring)
Time to transformation | From treatment start to transformation or progression without transformation or death or last follow-up, up to 13 years of follow-up
  Time elapsed between treatment start and transformation (event), progression without transformation (censoring), death (censoring) or last follow-up (censoring)

CONTACTS AND LOCATIONS:
Overall Officials: Davide Rossi, MD, PhD, Principal Investigator — Oncology Institute of Southern Switzerland
Locations (4):
- Italy (2):
  - Arcispedale Santa Maria Nuova, AUSL IRCSS, Hematology Department, Reggio Emilia, RE
  - Azienda Ospedaliera Universitaria Maggiore della Carità, Novara
- Switzerland (2):
  - Institute of Oncology Research, Bellinzona, Canton Ticino
  - Institute of Pathology, Locarno, Canton Ticino